CLINICAL TRIAL: NCT00305214
Title: Microvolt T Wave Alternans Testing for Risk Stratification of Post MI Patients (MASTER II)
Brief Title: MASTER II - Microvolt T Wave Alternans Testing for Risk Stratification of Post MI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Brett Peterson / Sr. Clinical Trial Leader, Medtronic CRDM Core Clinical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 220b
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Myocardial Infarction; Arrhythmia, Ventricular; Ischemic Cardiomyopathy
Keywords: Myocardial Infarction; Microvolt T Wave Alternans Test; Implantable Cardioverter Defibrillator (ICD); Ventricular Arrhythmia
MeSH Terms: conditions — Myocardial Infarction; Arrhythmias, Cardiac

INTERVENTIONS:
Procedure: T Wave Alternans Test

SUMMARY:
The purpose of the study is to determine the usefulness of Microvolt T Wave Alternans (MTWA) testing of patients that have had a heart attack and have decreased pumping ability of the lower chamber of their heart. MTWA testing is a non-invasive test used to detect the likelihood of developing abnormally fast rhythms in the lower chambers of the heart. The objective of the study is to prove that if a patient has a positive MTWA test, they will be more likely to develop abnormally fast and dangerous rhythms in the lower chambers of the heart. The results of the study will help doctors to determine which patients would benefit the most from having an Implantable Cardioverter Defibrillator (ICD) implanted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of heart attacks
* LVEF >0.30 and <= 0.40 as measured by a radionuclide study, angiography or quantitative echocardiography within 3 months prior to enrollment.

Exclusion Criteria:

* Patients with electrocardiographically documented sustained ventricular tachycardia, ventricular fibrillation or prior cardiac arrest (Class I indications)
* Patients who have undergone an electrophysiologic study with ventricular stimulation or a MTWA test within 1 year prior to enrollment
* Patients with medical conditions that preclude the testing required by the Investigational Plan or limit study participation
* Patients unable to complete MTWA testing requirements due to current atrial fibrillation or flutter
* Patients unable to exercise and for which alternative modalities (pacing or pharmacological stress) used for MTWA testing are not available
* Patients who have experienced an MI within 1 month prior to enrollment
* Patients with advanced cerebrovascular disease per physician's assessment
* Patients classified as NYHA Class IV at time of enrollment
* Patients who have undergone cardiac revascularization within 3 months prior to enrollment or are scheduled for cardiac revascularization at the time of enrollment
* Patients with a life expectancy of less than 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405
Dates: Start 2003-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the life-threatening ventricular tachyarrhythmic event-free survival probability is greater in patients with a baseline MTWA Negative result as compared to patients with a baseline MTWA Positive result.

SECONDARY OUTCOMES:
Compare occurrence of all ventricular events between both groups
Identify predictors of life threatening ventricular arrhythmias
Calculate occurrence of life threatening ventricular arrhythmias based on last MTWA results

CONTACTS AND LOCATIONS:
Overall Officials: David G. Benditt, MD, Study Chair — University of Minnesota; Theodore Chow, MD, Study Chair — The Lindner Center for Research and Education; Dean J. Kereiakes, MD, FACC, Study Chair — The Lindner Center for Research and Education
Locations (47):
- United States (47):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Walnut Creek, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Hollywood, Florida
  - Naples, Florida
  - Safety Harbor, Florida
  - Atlanta, Georgia
  - Joliet, Illinois
  - Springfield, Illinois
  - Beech Grove, Indiana
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Hyannis, Massachusetts
  - Grand Rapids, Michigan
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - East Islip, New York
  - Flushing, New York
  - West Islip, New York
  - Gastonia, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scranton, Pennsylvania
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Amarillo, Texas
  - Corpus Christi, Texas
  - Plano, Texas
  - Tyler, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Portsmouth, Virginia
  - Appleton, Wisconsin